CLINICAL TRIAL: NCT06633393
Title: Impact of Feedback Based on the Myopia Prediction System on High Myopia Risk and Consultation Behavior in School-aged Children: a Cluster Randomized Controlled Trial
Brief Title: Effect of a Myopia Prediction System on Myopia Prevention and Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Prof., Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024KYPJ102
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Myopia; Randomized Controlled Trials; Artificial Intelligence (AI)
Keywords: Myopia Prediction; Randomized Controlled Trials; Artificial Intelligence (AI)
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): At baseline and six months, feedback on ophthalmic examination results and future high myopia risk at 18 years of age using the myopia prediction system
  Interventions: Other: Feedback on Predicted High Myopia Risk at Age 18 Using the Myopia Prediction System; Other: Feedback on Ophthalmic Examinations
- Control Arm (Active Comparator): At baseline and six months, feedback on ophthalmic examination results.
  Interventions: Other: Feedback on Ophthalmic Examinations

INTERVENTIONS:
Other: Feedback on Predicted High Myopia Risk at Age 18 Using the Myopia Prediction System — At baseline and six months, participants will be provided with the results of their predicted risk of high myopia at age 18 based on the myopia prediction system.
  Arms: Experimental Arm
Other: Feedback on Ophthalmic Examinations — At baseline and six months, participants will be provided with the results of their ophthalmic examinations.

SUMMARY:
The global rise in myopia, particularly among children and adolescents in China, underscores the inadequacy of current prevention strategies, indicating that conventional screening and education alone are insufficient to curb the prevalence. Integrating personalized myopia prediction into routine care may enhance risk awareness, promote proactive prevention, and improve adherence to medical advice, ultimately reducing the future burden of high myopia.

A myopia prediction system based on artificial intelligence was previously developed, accurately predicting future high myopia risk using efficient, robust, and easily accessible predictive factors, including age, spherical equivalent, and the annual progression of spherical equivalent. This study aims to conduct a prospective, one-year, cluster randomized controlled clinical trial to investigate the effectiveness of this prediction system in preventing and controlling myopia in school-aged children.

ELIGIBILITY:
Inclusion Criteria:

* The participant and their guardian voluntarily signed the informed consent form
* Has the record of eye refraction examination in the past year
* Aged 9 to 11 years, regardless of gender

Exclusion Criteria:

* High myopia(spherical equivalent ≤ -6.00 D)
* Ocular diseases other than myopia (e.g., strabismus, amblyopia, congenital cataract, juvenile glaucoma, retinal diseases).
* Systemic diseases that may affect vision or visual development (e.g., diabetes or other endocrine disorders, cardiovascular or respiratory diseases, Down syndrome)

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20000 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of Individuals Predicted to Develop High Myopia at Age 18 by the Myopia Prediction System | 1 year
  At the end of the one-year study, the Myopia Prediction System will be used to predict whether students will develop high myopia at age 18 in both the intervention and control groups. The Proportion of Individuals Predicted to Develop High Myopia at Age 18 by the Myopia Prediction System is calculated as the total number of students in each group predicted to develop high myopia by age 18, divided by the total number of students in the respective group.
Cumulative Clinical Visit Rate for Myopia Prevention and Control | Within 3 months after each intervention
  The Cumulative Clinical Visit Rate Proportion of Clinical Visits for Myopia Prevention and Control is the proportion of students in the intervention or control group who visited a hospital or clinic for myopia-related care (e.g., refractive exams and treatment) at least once within three months of either intervention. It is calculated as the number of students in each group who attended a clinical visit within three months of at least one intervention, divided by the total number of students in the respective group.

SECONDARY OUTCOMES:
Myopia Incidence Rate | 1 year
  1-year myopia incidence rate = number of new myopia cases within one year / number of non-myopic cases at baseline * 100%
Changes in Spherical Equivalent | 1 year
  Change in spherical equivalent (non-cycloplegic autorefraction) will be calculated
Screen Time | 1 year
  Daily usage time of electronic devices (computer/smartphone/tablet computer) will be calculated
Outdoor Activity Time | 1 year
  Daily outdoor activity time will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin H, Long E, Ding X, Diao H, Chen Z, Liu R, Huang J, Cai J, Xu S, Zhang X, Wang D, Chen K, Yu T, Wu D, Zhao X, Liu Z, Wu X, Jiang Y, Yang X, Cui D, Liu W, Zheng Y, Luo L, Wang H, Chan CC, Morgan IG, He M, Liu Y. Prediction of myopia development among Chinese school-aged children using refraction data from electronic medical records: A retrospective, multicentre machine learning study. PLoS Med. 2018 Nov 6;15(11):e1002674. doi: 10.1371/journal.pmed.1002674. eCollection 2018 Nov. PMID 30399150